CLINICAL TRIAL: NCT07127549
Title: Assessment of Core Muscle Strength, Endurance, and Balance in Women With Urinary Incontinence
Brief Title: Core Muscle Strength, Endurance, and Balance in Women With Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: Seda Saka (Other)
Responsible Party: Sponsor-Investigator, Seda Saka, Principal investigator, PhD, PT, Halic University
Organization: Halic University (Other)
Other Study IDs: ssaka9
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; core strength; core endurance; balance
MeSH Terms: conditions — Urinary Incontinence | interventions — Muscle Strength

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Muscle strength, endurance and balance assessment — All participants were administered a demographic assessment form; the International Physical Activity Questionnaire-Short Form (IPAQ-SF) to assess physical activity level; the Pelvic Floor Distress Inventory (PFDI-20) and all of its subscales to evaluate the severity of symptoms associated with pelvic floor distress; urodynamic measurement; a pad test to assess the severity of UI; a perineometer device to evaluate pelvic floor muscle (PFM) strength; the Sahrmann five-level core stabilization test and the Stabilizer Pressure Biofeedback Unit to assess core muscle strength; McGill's Trunk Endurance Tests for core endurance; and the Y Balance Test to assess balance.

SUMMARY:
Urinary incontinence (UI) is defined as the involuntary loss of urine that occurs outside the individual's control and negatively affects both hygiene and social life. Research indicates that individuals with UI experience decreased core muscle strength and endurance, which may also lead to changes in balance parameters. Therefore, the aim of this study was to investigate core muscle strength, endurance, and balance parameters in women with UI, taking the type of UI into consideration.

This study was conducted between January 2025 and April 2025 at the Urogynecology Clinic of Başakşehir Çam and Sakura City Hospital in Istanbul, with patients diagnosed with UI by a specialist physician. A total of 32 participants were included. All participants were administered a demographic assessment form; the International Physical Activity Questionnaire-Short Form (IPAQ-SF) to assess physical activity level; the Pelvic Floor Distress Inventory (PFDI-20) and all of its subscales to evaluate the severity of symptoms associated with pelvic floor distress; urodynamic measurement; a pad test to assess the severity of UI; a perineometer device to evaluate pelvic floor muscle (PFM) strength; the Sahrmann five-level core stabilization test and the Stabilizer Pressure Biofeedback Unit to assess core muscle strength; McGill's Trunk Endurance Tests for core endurance; and the Y Balance Test to assess balance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with urinary incontinence by a specialist physician
* Native Turkish speaker
* Willing to participate in the study

Exclusion Criteria:

* Pregnant
* Given birth within the past year
* Cooperation problems
* Presence of urinary infection
* Diagnosed with pelvic organ prolapse (POP) stage higher than 2
* History of pelvic surgery
* Presence of dizziness, vertigo, tinnitus, hearing loss, or ear fullness (uncontrolled vestibulopathies)
* Use of medications that affect balance
* Resistance to digital vaginal palpation or insertion of a perineometer into the vagina
* Orthopedic, cognitive, cardiac, or neurological conditions that may prevent participation in the study

Ages: 35 Years to 55 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female
Study Population: All patients who applied to the Urogynecology Clinic at Başakşehir Çam and Sakura City Hospital and were diagnosed with urinary incontinence by a specialist physician constitute the population of the study. The sample of the study consists of 32 women from this population who met the inclusion and exclusion criteria and agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Assessment of Pelvic Floor Muscle Strength | At the day of enrollment
  a previously validated perineometer with good inter-rater reliability and reproducibility was used to assess pelvic floor muscle strength.
  a previously validated perineometer with good inter-rater reliability and reproducibility was used to assess pelvic floor muscle strength.
  A previously validated perineometer with good inter-rater reliability and reproducibility was used to assess pelvic floor muscle strength.
Assessment of Urine Flow Rate and Volume | At the day of enrollment
  A uroflowmetry device was used to assess urine flow rate and volume.
  A uroflowmetry device was used to assess urine flow rate and volume
Assessment of Urinary Incontinence Severity | At the day of enrollment
  A 1-hour pad test was used to determine the severity of urinary incontinence.
Assessment of Core Muscle Strength | At the day of enrollment
  The Stabilizer Pressure Biofeedback Unit® (Chattanooga Medical Supply Inc., Chattanooga, TN) was used to determine the level of core stabilization.
Assessment of Core Endurance and Stability | At the day of enrollment
  The test protocol developed by McGill and colleagues was applied to measure core endurance.
Balance Assessment | At the day of enrollment
  The Y Balance Test was used to assess balance.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | At the day of enrollment
  The IPAQ-SF is a brief self-report questionnaire used to assess the physical activity levels of individuals over the past 7 days. It measures the frequency and duration of walking, moderate-intensity, and vigorous-intensity activities.
Pelvic Floor Distress Inventory-20 (PFDI-20) | At the day of enrollment
  The PFDI-20 is a questionnaire designed to evaluate the presence and severity of pelvic floor distress symptoms, including urinary, colorectal, and pelvic organ prolapse symptoms. It helps assess the impact of these symptoms on a patient's quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided